CLINICAL TRIAL: NCT02856607
Title: Impact of Clinical Care Pathway on Prognosis and Therapeutic Medical Care of Infective Endocarditis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_3675
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Infective Endocarditis (IE)
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group I: patient for whom diagnosis and medical care are realized in a referent center with cardiac surgery
  Interventions: Other: determine the prognosis of threated patients according to the clinical care pathway.
- Group II: patients secondary addressed to a referent center with cardiac surgery
  Interventions: Other: determine the prognosis of threated patients according to the clinical care pathway.
- Group III: patients for which the totality medical care are performed in non-referent health center
  Interventions: Other: determine the prognosis of threated patients according to the clinical care pathway.

INTERVENTIONS:
Other: determine the prognosis of threated patients according to the clinical care pathway.

SUMMARY:
Infective endocarditis (IE) is defined as a bacterial infection of the endocardium (inner surface of the heart), which may include one or more heart valves. Epidemiologic pattern has changed during the last 20 years whereas the incidence was unchanged. However, the mortality increase despite recent diagnosis and therapeutic advances.

Only few investigations consider the prognostic and the therapeutic medical care according to the clinical care pathway. In fact, 3 situations are observed: (i) patient for whom diagnosis and medical care are realized in a referent center with cardiac surgery, (ii) patients secondary addressed to a referent center with cardiac surgery, (iii) patients for which the totality medical care are performed in non-referent health center. In addition, epidemiologic studies concern only a part of IE, not including most of the time the patients hospitalized in non-referent center.

The aim of the study was to determine the prognosis of threated patients according to the clinical care pathway. Secondary objectives was (i) to evaluate the application of European recommendations concerning trans-oesophageal echocardiogram (TOE), antibiotic treatment and surgical practice, (ii) to compare the epidemiologic profile according to the type of center.

For this, 300 patients addressed in the 22 French participating centers for a possible or certain IE according to Duke Criteria were prospectively included during 3 years.

Patient data (clinical, demographical, biological, microbiological, echocardiographic and evolutive data) were collected at the admission, during hospitalization, at discharge and one-year follow up.

ELIGIBILITY:
Inclusion Criteria:

- adult with infective endocarditis episode according to Duke Criteria

Exclusion Criteria:

* Patients with a new episode of infective endocarditis that led to its prior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adults with infective endocarditis episode
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the all-cause one-year mortality according to the group | one year

SECONDARY OUTCOMES:
the application of European recommendations | one year
  realization of trans-oesophageal echocardiogram (TOE)
antibiotic treatment | one year
  type and time of antibiotic treatment for common germ,
surgery | one year
  performing valve surgery and / or total extraction of an implanted pacemaker or defibrillator.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpoitaux de Marseille Hôpital de la Timone, Marseille, France